CLINICAL TRIAL: NCT06766981
Title: Effectiveness of Local Anesthetic Infiltration With Articaine 4% in Comparison to Inferior Alveolar Nerve Block With Lidocaine 2% for Mandibular 1st Molar Extraction
Brief Title: Infiltration Anesthesia vs. Block Anesthesia
Acronym: LAI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sinan A. Shwailiya (Other)
Collaborators: Babylon University (Other)
Responsible Party: Sponsor-Investigator, Sinan A. Shwailiya, Lect.Dr, Babylon University
Organization: Babylon University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 35/2024
Record Dates: First submitted 2025-01-04; First posted 2025-01-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-01

CONDITIONS: Tooth Extraction
Keywords: Local Anesthesia; Inferior Dental Nerve Block; Infiltration Anesthesia
MeSH Terms: interventions — Anesthesia, Conduction

STUDY DESIGN:
Intervention Model Description: The interventional group will undergo tooth extraction under the infiltration anaesthesia technique
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Block (Active Comparator): This group will receive a conventional inferior alveolar nerve block (IANB) technique with 2% lidocaine with epinephrine (1:80,000) for tooth extraction.
  Interventions: Procedure: Inferior Alveolar Nerve Block
- Infiltration (Experimental): This group will receive 4% articaine with 1:100,000 epinephrine as lingual and buccal infiltration for tooth extraction
  Interventions: Procedure: Infiltration with Articain 4%

INTERVENTIONS:
Procedure: Infiltration with Articain 4% — The experimental group of patients that are diagnosed for tooth extraction of mandibular 1st. molar will undergo extraction using an infiltration technique for local anaesthesia. In contrast to the conventional group that will receive Inferior alveolar nerve block
  Arms: Infiltration
Procedure: Inferior Alveolar Nerve Block — This group will receive a conventional inferior alveolar nerve block (IANB) technique with 2% lidocaine with epinephrine (1:80,000) for tooth extraction.
  Other Names: Regional Anaesthesia
  Arms: Block

SUMMARY:
Checking the effectiveness of the infiltration technique of local anesthetic agent as an alternative to inferior dental nerve block during tooth extraction

DETAILED DESCRIPTION:
Patients who need their Mandibular first Molar to be removed under local anaesthesia. The first group will receive 4% articaine with 1:100,000 epinephrine as lingual and buccal infiltration. In comparison, the second group will receive a conventional inferior alveolar nerve block technique with 2% lidocaine with epinephrine (1:80,000). Pain will be measured para-operatively using a verbal rating scale.

ELIGIBILITY:
Inclusion Criteria:

* The systemic condition must be normal.
* Patient has no cardiovascular, metabolic, or transmitted disease.
* The patient has a Mandibular 1st. Molar tooth indicated for extraction.
* The tooth is non-restorable.

Exclusion Criteria:

* Chronic cardiovascular condition, metabolic, or infectious disease.
* Pregnant women.
* The tooth is restorable.

Ages: 18 Years to 58 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-02-10 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Verbal Pain Rating Scale | during the intervention/procedure/surgery
  Pain during tooth extraction will be measured immediately after the procedure is completed using a verbal rating scale. The zero rate will be given when the patient feels no pain; the rating degree will increase as the pain severity becomes more severe. According to the following scale:
  0 No hurt
  1. Slight pain
  2. Moderate pain
  3. Intense pain
  4. Extremely painful

CONTACTS AND LOCATIONS:
Locations (2):
- Iraq (2):
  - College of Dentistry, University of Babylon, Hillah, Babylon
  - College of Dentistry/University of Babylon, Hillah, Babylon

IPD SHARING:
Plan to Share IPD: Yes
Study DATA will be provided on request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: after research publishment
Access Criteria: other researchers

REFERENCES:
- [Background] Bataineh AB, Nusair YM, Al-Rahahleh RQ. Comparative study of articaine and lidocaine without palatal injection for maxillary teeth extraction. Clin Oral Investig. 2019 Aug;23(8):3239-3248. doi: 10.1007/s00784-018-2738-x. Epub 2018 Nov 12. PMID 30417227
- [Background] Madden VJ, Kamerman P, Leake HB, Catley MJ, Heathcote LC, Moseley GL. The Sensation and Pain Rating Scale: easy to use, clear to interpret, and responsive to clinical change. medRxiv [Preprint]. 2024 Jan 9:2023.09.08.23295128. doi: 10.1101/2023.09.08.23295128. PMID 37732279